CLINICAL TRIAL: NCT00527410
Title: A Phase I Safety and Pharmacokinetic Study of Intravenous RTA 744 Injection in Patients With Recurrent, Progressive or Refractory Neoplastic Meningitis
Brief Title: A Safety Study of RTA 744 in Recurrent, Progressive or Refractory Neoplastic Meningitis
Acronym: LMD
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business Decision
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RTA 744-C-0601
Record Dates: First submitted 2007-09-07; First posted 2007-09-10 (Estimated); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Leptomeningeal Carcinomatosis
MeSH Terms: conditions — Meningeal Carcinomatosis | interventions — WP 744

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- RTA 744 (Experimental): RTA 744 injection administered intravenously for a maximum of 18 cycles (54 weeks). Dose escalation based on four dose levels and occurance of dose limiting toxicity (DLT).
  Interventions: Drug: RTA 744

INTERVENTIONS:
Drug: RTA 744 — Aqueous solution of RTA 744 is packaged in 5 ml vials - 1 mg/ ml. The drug is mixed in D10W and infused over 2 hours on three consecutive days.

SUMMARY:
This study assesses the tolerability, safety, efficacy and pharmacokinetics of RTA 744 in recurrent neoplastic meningitis.

DETAILED DESCRIPTION:
Neoplastic meningitis refers to the deposition of malignant cells in the lining (leptomeninges) of the brain and spine. Neoplastic meningitis from solid tumors most often occurs in patients with advanced systemic disease who have failed prior chemotherapy; it is also frequent in patients with CNS parenchymal metastasis. Patient survival remains low, and better treatments are needed to penetrate the blood brain barrier and treat the entire neuraxis.

RTA 744 is a close chemical analogue of the well characterized anti-cancer agent doxorubicin. Unlike doxorubicin, RTA 744 has shown ability to cross the blood brain barrier and to achieve high concentration in CNS tumor tissue in animal models. Dose escalation will continue as pre-determined until first occurrence of a dose-limiting toxicity. Maximum tolerated dose will be determined as defined in protocol.

ELIGIBILITY:
Inclusion Criteria:

* Histologic confirmation of primary malignancy. All primary tumor types may be enrolled.
* Neoplastic meningitis/leptomeningeal metastasis refractory to conventional therapy with presence of tumor cells on cytology, OR neuroimaging evidence of leptomeningeal tumor by MRI.
* Not eligible for higher priority clinical trial.
* Have recovered from side effects of any surgical resection.
* A stable dose of steroid for at least 7 days prior to the Gd-MRI.
* Karnofsky Performance Status (KPS) of ≥ 60.
* Laboratory Parameters: ANC ≥ 1.5 x 109/L; Hgb ≥ 9 g/dl; Platelets ≥ 100 x 109/L; AST and ALT ≤ 3.0 x ULN; Serum bilirubin ≤ 1.5 x ULN; Serum creatinine ≤ 1.5 x ULN; 24 hour creatinine clearance ≥ 50 ml/min
* Life expectancy of at least 8 weeks.
* Written informed consent obtained.

Exclusion Criteria:

* Concurrent therapy for leptomeningeal disease or other malignancy.
* Clinical evidence of obstructive hydrocephalus or compartmentalization of CSF flow.
* Cumulative doses: doxorubicin > 450 - 550 mg/m2, epirubicin > 800-1000 mg/m2, idarubicin >130-150 mg/m2 and daunorubicin > 400-550 mg/m2.
* Anticonvulsant medications or other types of medications which are known to induce the CYP450 enzymes.
* Pregnancy or breast feeding, or adults (male or female) of reproductive potential not employing an effective method of birth control
* Total 24 hour urinary protein > 500 mg.
* Concurrent severe and/or uncontrolled medical conditions which could compromise participation in the study
* Impaired cardiac function, other significant prior cardiac disease or arrhythmia of any type
* Myocardial infarction ≤ 6 months prior
* History of CHF or arrhythmias
* Therapeutic doses of anticoagulant therapy (prophylactic dosing is allowed)
* Investigational drugs less than 4 weeks prior; intrathecal chemotherapy within 2 weeks prior; systemic cytotoxic chemotherapy within 4 weeks prior (6 weeks for nitrosourea or mitomycin-C or 2 weeks for vincristine); radiation therapy within 2 weeks prior; any medication known to cause QT interval prolongation
* Any surgery <2 weeks prior

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2006-10-31 (Actual); Primary Completion 2008-12-01 (Actual)

PRIMARY OUTCOMES:
Determine the tolerability of RTA 744 Injection in patients with leptomeningeal disease (LMD) secondary to any type of primary tumor. | evaluation at end of cycle 1 for each cohort
Characterize the multiple-dose pharmacokinetics of RTA 744 in plasma and CSF in a selected group of 6-10 patients who will receive RTA 744 at or near the maximum tolerated dose (MTD). | end of study

SECONDARY OUTCOMES:
Document any potential antitumor activity. | after every even numbered treatment cycle
Correlate pharmacokinetic information with clinical (efficacy and safety) responses. | end of study

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/